CLINICAL TRIAL: NCT02939885
Title: Imagerie Fonctionnelle cérébrale: Aspects Normaux et Pathologiques
Brief Title: fMRI Study of Brain Mechanisms Related to Emotions
Acronym: ICF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other)
Responsible Party: Sponsor
Other Study IDs: P/2006/50
Record Dates: First submitted 2016-09-05; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to better define and understand the brain mechanisms related to emotional and cognitive dimensions using odorous stimuli, gustatory stimuli, visual stimuli and auditory stimuli using functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* Healthy Volunteers

Exclusion Criteria:

* those applied for an magnetic resonance examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants came after invitation to volunteer. They are mainly students from our university.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cerebral activation of subjects using Blood Oxygenation Level Dependant (BOLD) contrast imaging | at admission
  measure brain activity by the BOLD technical

REFERENCES:
- [Result] Bonnet L, Comte A, Tatu L, Millot JL, Moulin T, Medeiros de Bustos E. The role of the amygdala in the perception of positive emotions: an "intensity detector". Front Behav Neurosci. 2015 Jul 7;9:178. doi: 10.3389/fnbeh.2015.00178. eCollection 2015. PMID 26217205
- [Result] Comte A, Gabriel D, Pazart L, Magnin E, Cretin E, Haffen E, Moulin T, Aubry R. On the difficulty to communicate with fMRI-based protocols used to identify covert awareness. Neuroscience. 2015 Aug 6;300:448-59. doi: 10.1016/j.neuroscience.2015.05.059. Epub 2015 May 30. PMID 26033566
- [Result] Gabriel D, Henriques J, Comte A, Grigoryeva L, Ortega JP, Cretin E, Brunotte G, Haffen E, Moulin T, Aubry R, Pazart L. Substitute or complement? Defining the relative place of EEG and fMRI in the detection of voluntary brain reactions. Neuroscience. 2015 Apr 2;290:435-44. doi: 10.1016/j.neuroscience.2015.01.053. Epub 2015 Jan 30. PMID 25644421
- [Result] Pazart L, Comte A, Magnin E, Millot JL, Moulin T. An fMRI study on the influence of sommeliers' expertise on the integration of flavor. Front Behav Neurosci. 2014 Oct 16;8:358. doi: 10.3389/fnbeh.2014.00358. eCollection 2014. PMID 25360093
- [Result] Galliot E, Comte A, Magnin E, Tatu L, Moulin T, Millot JL. Effects of an ambient odor on brain activations during episodic retrieval of objects. Brain Imaging Behav. 2013 Jun;7(2):213-9. doi: 10.1007/s11682-012-9218-8. PMID 23292620
- [Result] Billot PE, Comte A, Galliot E, Andrieu P, Bonnans V, Tatu L, Gharbi T, Moulin T, Millot JL. Time course of odorant- and trigeminal-induced activation in the human brain: an event-related functional magnetic resonance imaging study. Neuroscience. 2011 Aug 25;189:370-6. doi: 10.1016/j.neuroscience.2011.05.035. Epub 2011 May 20. PMID 21620934
- [Result] Lombion S, Comte A, Tatu L, Brand G, Moulin T, Millot JL. Patterns of cerebral activation during olfactory and trigeminal stimulations. Hum Brain Mapp. 2009 Mar;30(3):821-8. doi: 10.1002/hbm.20548. PMID 18330871